CLINICAL TRIAL: NCT00720655
Title: Effects of Fatty and Lean Fish Intake on Cardiovascular Risk Factors in Subjects With Coronary Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Collaborators: Kuopio University Hospital (Other)
Responsible Party: Arja Erkkilä, University of Kuopio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FISH6417
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Blood Pressure; Arrhythmia; Inflammation
Keywords: coronary heart disease
MeSH Terms: conditions — Arrhythmias, Cardiac; Inflammation; Coronary Disease | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fatty fish (Experimental)
  Interventions: Other: Dietary intervention
- Lean Fish (Experimental)
  Interventions: Other: Dietary intervention
- Control diet (Placebo Comparator)
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — Fatty fish at least 4 meals per week.
  Arms: Fatty fish
Other: Dietary intervention — Lean fish at least 4 meals per week.
  Arms: Lean Fish
Other: Dietary intervention — Control diet with lean meat and chicken.
  Arms: Control diet

SUMMARY:
The aim of the study is to examine the effects of fatty fish and white (lean) fish on cardiovascular disease risk factor levels in subjects with established coronary heart disease using multiple medications. The main end points are blood pressure, serum lipids, inflammatory markers, arrhythmias and gene expression in peripheral mononuclear cells. The study design was a controlled, parallel study lasting 8 weeks with three diet groups: fatty fish, white fish and control group (lean pork, beef or chicken).

ELIGIBILITY:
Inclusion Criteria:

* myocardial infarction or unstable ischemic attack
* use of beta blockers
* normal sinus rhythm
* fasting serum triglyceride less or equal to 3.5 mmol/l
* fasting serum cholesterol less or equal to 8 mmol/l
* BMI 18.5-30 kg/m2
* fasting plasma glucose less or equal to 7 mmol/l

Exclusion Criteria:

* diabetes
* use of other antiarrhythmic medications than beta blockers
* atrial fibrillation
* use of psychotropic medications
* abnormal liver, thyroid or kidney function
* inflammatory bowel disease
* excessive use of alcohol
* use of fish oil supplements or high habitual intake of fish

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2005-08; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
gene expression in peripheral mononuclear blood cells, risk of arrhythmias, serum lipids and blood pressure | 8 week

SECONDARY OUTCOMES:
inflammatory markers | 8 week

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kuopio, Kuopio, Finland

REFERENCES:
- [Result] Erkkila AT, Schwab US, de Mello VD, Lappalainen T, Mussalo H, Lehto S, Kemi V, Lamberg-Allardt C, Uusitupa MI. Effects of fatty and lean fish intake on blood pressure in subjects with coronary heart disease using multiple medications. Eur J Nutr. 2008 Sep;47(6):319-28. doi: 10.1007/s00394-008-0728-5. Epub 2008 Jul 29. PMID 18665413
- [Derived] de Mello VD, Lankinen M, Schwab U, Kolehmainen M, Lehto S, Seppanen-Laakso T, Oresic M, Pulkkinen L, Uusitupa M, Erkkila AT. Link between plasma ceramides, inflammation and insulin resistance: association with serum IL-6 concentration in patients with coronary heart disease. Diabetologia. 2009 Dec;52(12):2612-5. doi: 10.1007/s00125-009-1482-9. Epub 2009 Aug 11. PMID 19669729
- [Derived] Lankinen M, Schwab U, Erkkila A, Seppanen-Laakso T, Hannila ML, Mussalo H, Lehto S, Uusitupa M, Gylling H, Oresic M. Fatty fish intake decreases lipids related to inflammation and insulin signaling--a lipidomics approach. PLoS One. 2009;4(4):e5258. doi: 10.1371/journal.pone.0005258. Epub 2009 Apr 23. PMID 19390588